CLINICAL TRIAL: NCT00477854
Title: Effects of Chromium Picolinate on Food Intake, Satiety, and Eating Attitudes in Overweight Women With Food Cravings
Brief Title: Effects of Chromium Picolinate on Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Nutrition 21, Inc. (Industry)
Responsible Party: Principal Investigator, William Cefalu, MD, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 24040
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Obesity; Atypical Depression
MeSH Terms: conditions — Obesity | interventions — picolinic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visual Analogue Scale Ratings (Experimental): Food intake data and its coefficients, including total food intake, food not eaten, duration of the meal, and bite rate. A mixed model analysis of variance will also be conducted on ratings of food cravings and eating atttudes. Changes in hunger and satiety ratings between, before, and after the meals will be compared for difference across treatment conditions.
  Interventions: Drug: Chromium Picolinate
- Consuming less Lunch allows consumption of more dinner (Experimental): Test whether chromium picolinate supplementation affects food cravings, eating attitudes, and satiety in healthy, overweight and/or obese, adult women who are determinded to be carbohydrate cravers. Whether participants who eat less at a lunch test meal consume more food at an ad lib dinner test meal with a diversity of foods.
  Interventions: Drug: Chromium Picolinate

INTERVENTIONS:
Drug: Chromium Picolinate — Test whether Chromium Picolinate supplementation affects food intake at both a test lunch meal and at a test dinner meal presented 4.5 hours later among healthy, overweight and/or obese, adult women who are determined to be carbohydrate creavers.

SUMMARY:
The purpose of this study is to test the effects of chromium picolinate on food intake, food cravings, eating attitudes, and appetite. If chromium picolinate is found to have a beneficial impact on satiety and food intake, then this supplement may be an alternative or adjunctive treatment for overweight people desiring to modify their food intake. The primary hypothesis of this study is that among individuals who report being carbohydrate cravers, chromium picolinate supplementation will reduce food intake during a test lunch meal and produce greater satiety in comparison to a placebo.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are:

1. Healthy female who has not been diagnosed with diabetes, cardiovascular illness, or other chronic diseases,
2. Food craver, determined by self-reported craving for carbohydrates on two out of three validated measures of food cravings,
3. > 18 years of age and < 50 years of age, and
4. Body mass index between 25 and 39.9 kg/m2. Participants will be scheduled for testing during the luteal phase of their menstrual cycle to limit the confounding effect of the menstrual cycle on energy intake. We will include women who are taking monophasic oral contraceptives but will exclude other oral contraceptive regimens. Participants with very irregular menstrual cycles will also be excluded because this irregularity will make it very difficult to schedule testing during the luteal phase of the menstrual cycle.

Exclusion Criteria:

Potential participants will be excluded for the following reasons:

1. Participants who report smoking cigarettes will be excluded because of the effects of nicotine upon taste and appetite,
2. Participants who have a diagnosable eating disorder (i.e., anorexia or bulimia nervosa) will also be excluded since intentional restriction of eating and binge eating/overeating could increase the variability of the data,
3. Participants who report using diet pills will be excluded since diet pills may potentially influence appetite, hunger, and/or satiety,
4. Participants will be excluded if they are taking anti-depressant medications, anti-psychotic medications, or any medications that may potentially influence appetite, hunger, and/or satiety,
5. Participants who are not determined to be carbohydrate cravers will be excluded,
6. Participants will also be excluded if they report any allergies to the foods that will be used in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2005-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Food intake at both a test lunch meal and at a test dinner meal presented 4.5 hours later | 8 weeks

SECONDARY OUTCOMES:
Hunger and satiety between the lunch and dinner meal | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Anton, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States